CLINICAL TRIAL: NCT03908775
Title: A Comparison of C-MAC Videolaryngoscopy and Direct Laryngoscopy for Nasotracheal Intubation in Children: A Randomized, Controlled Clinical Trial
Brief Title: A Comparison of C-MAC Videolaryngoscopy and Direct Laryngoscopy for Nasotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ülkü Özgül, Associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: UlkuNT
Record Dates: First submitted 2019-04-08; First posted 2019-04-09 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Intubation; Videolaryngoscopy; Children
Keywords: Intubation; Children; Hemodynamics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group VL (Active Comparator): C-MAC Videolaryngoscope Patients intubated with C-MAC Videolaryngoscope
  Interventions: Device: C-MAC videolaryngoscope
- Group DL (Active Comparator): Direct Laryngoscope Patients intubated with Direct laryngoscope
  Interventions: Device: Direct Laryngoscope

INTERVENTIONS:
Device: C-MAC videolaryngoscope — An intubating device that is used for nasotracheal intubation in children undergoing dental interventions. Nasotracheal intubation was applied by anesthesiologist with C-MAC videolaryngoscope.
  Arms: Group VL
Device: Direct Laryngoscope — An intubating device that is used for nasotracheal intubation. Nasotracheal intubation was applied by anesthesiologist with direct laryngoscope.
  Arms: Group DL

SUMMARY:
Nasotracheal intubation is indicated in patients undergoing oral, maxillofacial, or dental procedures. During nasal intubation with the traditional Macintosh laryngoscope, use of Magill's forceps or external laryngeal manipulation is usually required to facilitate intubation. The prolonged or multiple intubation attempts and, subsequently, may be associated with complications such as oxygen desaturation or airway and dental injuries.

The C-MAC videolaryngoscope (Karl Storz, Tuttlingen, Germany) is a videolaryngoscope using a modified Macintosh blade, which may be a useful alternative both for routine and difficult airway management and for educational purposes.

In this prospective, randomized, controlled trial, the purpose is to compare C-MAC and DL in terms of intubation times, hemodynamic response and adverse events associated with nasotracheal intubation in children undergoing dental procedures.

DETAILED DESCRIPTION:
Tracheal intubation using direct laryngoscopy is successful in the majority of patients, even when a line-of-sight view of the glottis is not possible. Although poor glottic visualization is encountered between 1% and 9% of attempts, success can generally be achieved with additional force, external laryngeal manipulation, or the use of gum elastic bougies and stylets. However, poor glottic exposure is more likely to require prolonged or multiple intubation attempts and, subsequently, may be associated with complications such as oxygen desaturation or airway and dental injuries. In recent years, videolaryngoscopy has begun to play an important role in the management of patients with an unanticipated difficult or failed laryngoscopic intubation.

The C-MAC videolaryngoscope (Karl Storz, Tuttlingen, Germany) is a videolaryngoscope using a modified Macintosh blade, which may be a useful alternative both for routine and difficult airway management and for educational purposes.

In this prospective, randomized, controlled trial, the purpose is to compare C-MAC and DL in terms of intubation times, hemodynamic response and adverse events associated with nasotracheal intubation in children undergoing dental procedures.

ELIGIBILITY:
Inclusion Criteria:

* 3-12 years
* American Society of Anesthesiology score I-II,
* undergoing dental procedure
* required nasotracheal intubation

Exclusion Criteria:

* Patients for risk of aspiration
* Upper airway abnormalities
* Known difficult airways

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Time to intubation | From beginning of inserting nasotracheal tube into nares to seeing two meaningful end-tidal carbon dioxide levels up to 3 minutes
  Time to intubation was defined as the time the nasotracheal tube was inserted into nares the until endtidal CO2 was detected

SECONDARY OUTCOMES:
Heart Rate | From beginning of Anesthesia induction to 10th minutes of intubation
  Heart Rate
Mean Arterial Pressure | From beginning of Anesthesia induction to 10th minutes of intubation
  Mean Arterial Pressure
Adverse Events | During the first 1 hour postoperatively
  Bleeding in the mouth and nose, the Magill Forceps use, burst of intubation tube cuff, external laryngeal pressure, presence of head position change, laryngospasm, hypoxia.

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Ozgul, Principal Investigator — Inonu University Faculty of Medicine
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim HJ, Kim JT, Kim HS, Kim CS, Kim SD. A comparison of GlideScope((R)) videolaryngoscopy and direct laryngoscopy for nasotracheal intubation in children. Paediatr Anaesth. 2011 Apr;21(4):417-21. doi: 10.1111/j.1460-9592.2010.03517.x. Epub 2011 Jan 19. PMID 21244568